CLINICAL TRIAL: NCT05174143
Title: Personalized Antiplatelet Therapy According to CYP2C19 Genotype in Coronary Artery Disease: A Real World Study
Brief Title: Personalized Antiplatelet Therapy in CAD Patients
Status: Completed | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Professor, Xinjiang Medical University
Other Study IDs: Y101310008
Record Dates: First submitted 2021-12-14; First posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Disease
Keywords: CYP2C19
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, no-randomized, single-center study performed on 15000 consecutive coronary artery patients from Dec. 2016 to Oct. 2021. All these patients were detected CYP2C19 genotype. The antiplatelet treatment was recorded according to the therapy actually adopted by the patients.

ELIGIBILITY:
Inclusion Criteria:

1.Aged >18 years old; 2. Coronary angiography confirmed that there was at least one coronary artery stenosis >70%; or the degree of stenosis of the left main artery stenosis >50%; 3. At least one clinical phenotype of coronary heart disease is present: stable angina or acute coronary syndrome 4.To be able to sign informed consent.

Exclusion Criteria:

1. Combined with severe valvular heart disease;
2. Combined with severe congenital heart disease;
3. Combined hyperthyroidism, anemia and other high-powered heart disease; 4. With pulmonary heart disease;

5. With hypertrophic obstructive cardiomyopathy; 6. Severe hypotension (SBP <90mmHg or DBP <60mmHg at enrollment); 7. Liver dysfunction (defined as ALT or total bilirubin is greater than the normal upper limit of 3 times); 8. Renal insufficiency (defined as serum creatinine greater than 1.5 times the normal upper limit); 9. High-risk bleeding patients, such as thrombocytopenia, blood diseases and other diseases; 10. active peptic ulcer and skin ulcers; 11. A patient who is allergic to clopidogrel, Ticagrelor, or aspirin; 12. Patients with a history of cardiogenic shock within two weeks; 13. pregnant and lactating women, during treatment can not be strict contraception of women of childbearing age; 14. In the past 3 months participated in other clinical researchers; 15. Persons who do not have legal or legal competence; 16. Any condition that the investigator considers unsuitable for participation in the clinical study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were ≥18 years of age, and coronary angiography confirmed that at least one coronary artery stenosis was ≥ 70% or that the left main stenosis was ≥50% amenable to PCI.
Sampling Method: Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Mortality | 5 years
  All-cause death and cardiac death
Net clinical adverse events | 5 years
  a composite of cardiac death, myocardial infarction (MI), revascularization, and bleeding (Bleeding Academic Research Consortium (BARC) definitions, type 2, 3, or 5),
bleeding events | 5 years
  BARC class 2 or higher bleeding events

SECONDARY OUTCOMES:
all-cause death | 5 years
  all-cause death
cardiac death | 5 years
  death for cardiac cause
stent thrombosis | 5 years
  according to the Academic Research Consortium criteria
myocardial infarction | 5 years
  defined in accordance with the universal definition proposed in 2007
stroke | 5 years
  including ischemic stroke and hemorrhage
urgent revascularization | 5 years
  with persistent or increasing symptoms need to intervention
major adverse cardiovascular events (MACE) | 5 years
  defined as cardiac death, cardiac death, MI, stent thrombosis, or urgent revascularization
major adverse cardiovascular and cerebrovascular events (MACCE) | 5 years
  cardiac death, stroke, MI, stent thrombosis, or urgent revascularization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu TT, Pan Y, Zheng YY, Wang ZL, Deng CJ, Wang S, Xie X. The U -shape relationship between free fatty acid level and adverse outcomes in coronary artery disease patients with hypertension: evidence from a large prospective cohort study. Lipids Health Dis. 2024 Sep 10;23(1):291. doi: 10.1186/s12944-024-02273-z. PMID 39256835
- [Derived] Wang SF, Wu TT, Zheng YY, Hou XG, Yang HT, Yang Y, Xie X. Serum Globulin to Albumin Ratio as a Novel Predictor of Adverse Clinical Outcomes in Coronary Artery Disease Patients Who Underwent PCI. Rev Cardiovasc Med. 2023 Oct 7;24(10):278. doi: 10.31083/j.rcm2410278. eCollection 2023 Oct. PMID 39077558
- [Derived] Pan Y, Wu TT, Deng CJ, Jiang ZH, Yang Y, Hou XG, Yan T, Wang S, Feng YJ, Zheng YY, Xie X. Association between the C-Reactive Protein-Albumin-Lymphocyte (CALLY) Index and Adverse Clinical Outcomes in CAD Patients after PCI: Findings of a Real-World Study. Rev Cardiovasc Med. 2024 Mar 25;25(4):111. doi: 10.31083/j.rcm2504111. eCollection 2024 Apr. PMID 39076545
- [Derived] Ning Y, Wang KY, Min X, Hou XG, Wu TT, Ma YT, Xie X. Cystatin C to Left Ventricular Ejection Fraction Ratio as a Novel Predictor of Adverse Outcomes in Patients with Coronary Artery Disease: A Prospective Cohort Study. Rev Cardiovasc Med. 2023 Sep 18;24(9):260. doi: 10.31083/j.rcm2409260. eCollection 2023 Sep. PMID 39076386
- [Derived] Wu TT, Pan Y, Zhi XY, Deng CJ, Wang S, Guo XX, Hou XG, Yang Y, Zheng YY, Xie X. Association between extremely high prognostic nutritional index and all-cause mortality in patients with coronary artery disease: secondary analysis of a prospective cohort study in China. BMJ Open. 2024 Jun 16;14(6):e079954. doi: 10.1136/bmjopen-2023-079954. PMID 38885991